CLINICAL TRIAL: NCT04708171
Title: The PROGRAM-study: Awake Mapping Versus Asleep Mapping Versus No Mapping for Glioblastoma Resections
Acronym: PROGRAM
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); Universitaire Ziekenhuizen KU Leuven (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jasper Gerritsen, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2020-081-2
Record Dates: First submitted 2020-11-26; First posted 2021-01-13 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Awake mapping under local anesthesia
  Interventions: Procedure: Awake mapping under local anesthesia
- Asleep mapping under general anesthesia
  Interventions: Procedure: Asleep mapping under general anesthesia
- Resection under general anesthesia without mapping
  Interventions: Procedure: Resection under general anesthesia without mapping

INTERVENTIONS:
Procedure: Awake mapping under local anesthesia — During an awake craniotomy, the patient is awake and cooperative during the resection of the tumor while the surgeon uses electro(sub)cortical mapping to prevent damage to eloquent areas.
  Groups: Awake mapping under local anesthesia
Procedure: Asleep mapping under general anesthesia — During asleep mapping under general anesthesia, the surgeon uses electro(sub)cortical mapping with evoked potentials (MEPs, SSEPs or continuous dynamic mapping) to prevent damage to eloquent areas.
  Groups: Asleep mapping under general anesthesia
Procedure: Resection under general anesthesia without mapping — During resection under general anesthesia without mapping, the surgeon does not use any intraoperative stimulation mapping techniques to identify eloquent areas.
  Groups: Resection under general anesthesia without mapping

SUMMARY:
The study is designed as an international, multicenter prospective cohort study. Patients with presumed glioblastoma (GBM) in- or near eloquent areas on diagnostic MRI will be selected by neurosurgeons. Patients will be treated following one of three study arms: 1) a craniotomy where the resection boundaries for motor or language functions will be identified by the "awake" mapping technique (awake craniotomy, AC); 2) a craniotomy where the resection boundaries for motor functions will be identified by "asleep" mapping techniques (MEPs, SSEPs, continuous dynamic mapping); 3) a craniotomy where the resection boundaries will not be identified by any mapping technique ("no mapping group"). All patients will receive follow-up according to standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤ 90 years
2. Tumor diagnosed as GBM on MRI as assessed by the neurosurgeon
3. Tumors situated in or near eloquent areas; motor cortex, sensory cortex, subcortical pyramidal tract, speech areas or visual areas as indicated on MRI (Sawaya Grading II and II)
4. The tumor is suitable for resection (according to neurosurgeon)
5. Written informed consent

Exclusion Criteria:

1. Tumors of the cerebellum, brain stem or midline
2. Multifocal contrast enhancing lesions
3. Medical reasons precluding MRI (e.g. pacemaker)
4. Inability to give written informed consent (e.g. because of severe language barrier)
5. Second primary malignancy within the past 5 years with the exception of adequately treated in situ carcinoma of any organ or basal cell carcinoma of the skin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with primary or recurrent glioblastoma (GBM).
Sampling Method: Probability Sample
Enrollment: 453 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Neurological morbidity | Between baseline and 6 weeks/3 months/6 months postoperatively
  NIHSS deterioration of 1 point or more as compared to baseline value.
Extent of resection | Assessed within 72 hours on postoperative MRI scan
  Resection percentage as assessed by an independent neuroradiologist on MRI contrast images with volumetric analysis

SECONDARY OUTCOMES:
Progression-free survival | Between surgery and 12 months postoperatively
  Progression-free survival (PFS) defined as time from diagnosis to disease progression (occurrence of a new tumour lesion with a volume greater than 0.175 cm³, or an increase in residual tumour volume of more than 25%) or death, whichever comes first.
Overall survival | Between surgery and 12 months postoperatively
  Overall survival (OS) defined as time from diagnosis to death from any cause.
Onco-functional outcome | Between baseline and 6 weeks/3 months/6 months postoperatively
  2D coordinate based on extent of resection (or residual tumor volume) on the x-axis and NIHSS score on the y-axis
Frequency and severity of Serious Adverse Events (SAEs) | Between surgery and 6 weeks postoperatively
  Infections, intracerebral bleeding, epilepsy, aphasia, paresis/paralysis in arms or/and legs (this is not an exhaustive list).
Residual tumor volume | Assessed within 72 hours on postoperative MRI scan
  Postoperative tumor volume in mm3 as assessed by an independent neuroradiologist on MRI contrast images with volumetric analysis
MRC deterioration (for motor gliomas) | Between baseline and 6 weeks/3 months/6 months postoperatively
  MRC deterioration of 1 point or more as compared to baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Gerritsen, MD, Study Director — Erasmus Medical Center
Locations (8):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium
- Germany (2):
  - University Hospital Heidelberg, Heidelberg
  - Technical University Munich, Munich
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Medical Center Haaglanden, The Hague, South Holland
- Inselspital Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerritsen JKW, Zwarthoed RH, Kilgallon JL, Nawabi NL, Jessurun CAC, Versyck G, Pruijn KP, Fisher FL, Lariviere E, Solie L, Mekary RA, Satoer DD, Schouten JW, Bos EM, Kloet A, Nandoe Tewarie R, Smith TR, Dirven CMF, De Vleeschouwer S, Broekman MLD, Vincent AJPE. Effect of awake craniotomy in glioblastoma in eloquent areas (GLIOMAP): a propensity score-matched analysis of an international, multicentre, cohort study. Lancet Oncol. 2022 Jun;23(6):802-817. doi: 10.1016/S1470-2045(22)00213-3. Epub 2022 May 12. PMID 35569489
- [Derived] Gerritsen JKW, Dirven CMF, De Vleeschouwer S, Schucht P, Jungk C, Krieg SM, Nahed BV, Berger MS, Broekman MLD, Vincent AJPE. The PROGRAM study: awake mapping versus asleep mapping versus no mapping for high-grade glioma resections: study protocol for an international multicenter prospective three-arm cohort study. BMJ Open. 2021 Jul 21;11(7):e047306. doi: 10.1136/bmjopen-2020-047306. PMID 34290067